CLINICAL TRIAL: NCT00584610
Title: The Effect of a Levonorgestrel-releasing Intrauterine Device Versus a Copper Containing Intrauterine Device on Coagulation Parameters
Brief Title: The Effect of a Levonorgestrel-releasing Intrauterine Device (IUD) Versus a Copper Containing IUD on Risk of Blood Clots
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vermont (Other)
Responsible Party: Kristen Wright, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 07-211
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Last update posted 2010-01-18 (Estimated); Status verified 2010-01

CONDITIONS: Blood Coagulation Disorders
Keywords: Women's health
MeSH Terms: conditions — Blood Coagulation Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Levonorgestrel-containing intrauterine device insertion
  Interventions: Device: Levonorgestrel-containing IUD (Mirena®)
- 2 (Active Comparator): Copper containing intrauterine device
  Interventions: Device: Copper-containing IUD (Paraguard®)

INTERVENTIONS:
Device: Levonorgestrel-containing IUD (Mirena®) — Levonorgestrel-containing intrauterine device insertion
  Other Names: Mirena
  Arms: 1
Device: Copper-containing IUD (Paraguard®) — Copper-containing intrauterine device insertion
  Other Names: Paraguard
  Arms: 2

SUMMARY:
This is a randomized controlled trial to assess the effect of a levonorgesterel-releasing intrauterine device (LNG IUD, Mirena®) versus a copper IUD (Paraguard®) on coagulation parameters known to be associated with risk of thrombosis (blood clots). Both the LNG IUD and the copper IUD are FDA approved devices for contraception.

Women enrolled in this study will be randomized to receive either the LNG IUD or the copper IUD. They will complete a one month bleeding diary prior to insertion of the IUD and again for one month while the IUD is in place. They will undergo phlebotomy (blood draw) at baseline (prior to insertion of the IUD), two and four months. Stored samples will be used to measure D-dimer, C-reactive protein (CRP), antithrombin (AT), factor VIIIc, activated partial thromboplastin time (aPTT) and activated partial thromboplastin time plus activated protein C (aPTT + APC). Both groups will undergo a GYN exam with screening for bacterial vaginosis and gonorrhea/chlamydia cultures prior to insertion of the IUD. A brief survey to assess the women's experience with the IUD, including symptomatology and satisfaction with the device, will be conducted at the four months after insertion.

ELIGIBILITY:
Inclusion Criteria:

* Women who desire long-term, reversible contraception

Exclusion Criteria:

* Women with coagulopathies
* History of thrombotic events
* Pregnancy
* Active pelvic infection
* Known hypersensitivity to progestin
* Undiagnosed vaginal bleeding
* Wilson's disease
* Sensitivity to copper
* Uterine anatomy that precludes insertion of an IUD
* Women with multiple sexual partners and history within the last 5 years of alcoholism or drug abuse.
* Additionally, women must be greater than 3 months postpartum and have had two months without oral contraceptive pills or 6 months without Depo Provera prior to enrollment.

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-12; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
The primary outcome of this study will be change in coagulation parameters, with sample size calculations powered to detect a 35% change in D-dimer within groups and a 50% difference between groups. | 4 years

SECONDARY OUTCOMES:
Patient satisfaction with IUD device | 4 years
Difference in bleeding patterns between groups | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Kristen P Wright, MD, Principal Investigator — University of Vermont; Julia V. Johnson, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Vermont, Burlington, Vermont, United States